CLINICAL TRIAL: NCT04279067
Title: Brain Computer Interface - Functional Electrical Stimulation (BCI-FES) Therapy for Stroke Rehabilitation
Brief Title: BCI-FES Therapy for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, An Do, Assistant Clinical Professor, Department of Neurology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20194936
Record Dates: First submitted 2020-02-12; First posted 2020-02-20 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: stroke
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The study is design as an early Phase II two-arm randomized trial. The experimental group will receive BCI-FES dorsiflexion therapy paired with conventional physiotherapy (Group 1), while the control arm will receive dose- and intensity-matched conventional physiotherapy (Group 2). A total of 80 chronic stroke survivors with gait impairment due to foot-drop will be recruited and randomized evenly into the 2 groups (33/group).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blinded to the whether participants are in Group 1 or 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BCI-FES dorsiflexion therapy with physiotherapy (Experimental): Subjects will undergo placement of an EEG cap using standard technique connected to our custom BCI system. Subjects will provide 5 min of training EEG data as they engage in alternating epochs of idling and attempted foot dorsiflexion (of the paretic side). In the online phase, the subjects will perform 20-25 BCI-FES runs. A total of 12 sessions will be performed at a rate of 3x/week (over 4 weeks). Each BCI-FES therapy session will be followed by 1 hour of conventional physiotherapy.
  Conventional Physical Therapy: This will consist of a standardized regimen of activities typical of conventional post-stroke gait therapy, including passive/active range of motion exercises (to reduce/prevent excessive plantarflexor contractures), lower-extremity muscle strengthening, and a progression from treadmill to overground walking exercises.
  Interventions: Device: BCI-FES dorsiflexion therapy; Behavioral: Physiotherapy one hour
- Dose-and intensity-matched physiotherapy (Experimental): Conventional Physical Therapy: This will consist of a standardized regimen of activities typical of conventional post-stroke gait therapy, including passive/active range of motion exercises (to reduce/prevent excessive plantarflexor contractures), lower-extremity muscle strengthening, and a progression from treadmill to overground walking exercises. A total of 12 sessions will be performed at 3x/week.
  In the dose-matched control group (Group 2), it will be 2 hours/session.
  Interventions: Behavioral: Physiotherapy two hours

INTERVENTIONS:
Device: BCI-FES dorsiflexion therapy — BCI technology enables "direct brain control" of external devices such as assistive devices and prostheses by translating brain waves into control signals. When BCI systems are integrated with functional electrical stimulation (FES) systems, they can be used to deliver a novel physical therapy to improve movement after stroke. The automated software will analyze the data to generate and calibrate a BCI decoder. In the online phase, the subjects will perform 20-25 BCI-FES runs. In each run, subjects will follow 10 alternating epochs of 10-s long idling/dorsiflexion textual cues, and respond by either idling or attempting dorsiflexion to elicit BCI-FES mediated contractions of the TA muscle.
  Arms: BCI-FES dorsiflexion therapy with physiotherapy
Behavioral: Physiotherapy one hour — This will consist of a standardized regimen of activities typical of conventional post-stroke gait therapy, including passive/active range of motion exercises (to reduce/prevent excessive plantarflexor contractures), lower-extremity muscle strengthening, and a progression from treadmill to overground walking exercises. A total of 12 sessions will be performed at 3x/week.
  Arms: BCI-FES dorsiflexion therapy with physiotherapy
Behavioral: Physiotherapy two hours — This will consist of a standardized regimen of activities typical of conventional post-stroke gait therapy, including passive/active range of motion exercises (to reduce/prevent excessive plantarflexor contractures), lower-extremity muscle strengthening, and a progression from treadmill to overground walking exercises. A total of 12 sessions will be performed at 3x/week.
  Arms: Dose-and intensity-matched physiotherapy

SUMMARY:
There are over 7 million stroke survivors in the US alone, with approximately 795,000 new cases annually. Despite the best available physiotherapy, 30-60% of stroke survivors remain affected by difficulty walking, with foot weakness often being the main cause. Given that post-stroke gait impairments remain poorly addressed, new methods that can provide lasting improvements are necessary. Brain-computer interface (BCI) technology may be one such novel approach. BCI technology enables "direct brain control" of external devices such as assistive devices and prostheses by translating brain waves into control signals. When BCI systems are integrated with functional electrical stimulation (FES) systems, they can be used to deliver a novel physical therapy to improve movement after stroke. BCI-FES systems are hypothesized to stimulate recovery after stroke beyond that of conventional physical therapy.

DETAILED DESCRIPTION:
Preliminary research indicates that applying this technique to foot weakness after stroke is safe and may improve walking function. Hence, this warrants further investigation to: 1. determine if BCI-FES therapy can provide lasting gains in walking in chronic stroke patients; 2. determine what factors influence BCI-FES therapy; and 3. explicitly elucidate the underlying neural repair mechanisms. First, a Phase II clinical trial in patients with foot drop due to chronic stroke will compare the effect of BCIFES dorsiflexion therapy to that of dose- and intensity-matched standard physical therapy (Aim 1). Comparing the improvement in walking speed and other secondary outcome measures between the two groups will test if BCI-FES therapy provides functional and neurological gains beyond those of standard physical therapy. The relationship between the patient baseline characteristics (walking speed, ankle function, stimulated muscle responses, brain wave features, sensation) and the outcomes will determine what features influence responsiveness to BCI-FES dorsiflexion therapy (Aim 2). Finally, the underlying mechanism driving the improvements of BCI-FES will be studied (Aim 3). Determining that BCI-FES therapy can provide improvements beyond that of standard therapy may lead to a new treatment for stroke patients. The underlying mechanism can inform the design of future physical therapy techniques or improve current ones. Finally, BCI-FES therapy may ultimately become a novel form of physical therapy to reduce post-stroke disability, and in turn reduce the public health burden of stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-80 years inclusively at time of consent;
2. Radiologically confirmed stroke, ischemic or intracerebral hemorrhage (ICH) in etiology, with day of onset at least 26 weeks prior to day of randomization
3. Gait velocity<0.8 m/s at screening and baseline visits.
4. Foot-drop in affected limb as defined by dorsiflexion active range of motion (AROM) via goniometry in seated position foot dangling is less than passive range of motion and less than 15 degrees.
5. Plantarflexors spasticity<3 on modified Ashworth Scale;
6. Can walk >10 m (with or without ankle foot orthosis (AFO), and cane or walker permitted) at a supervised level;
7. Can tolerate FES with pain no more than 4 on pain analog scale and has adequate muscle response of dorsiflexion ≥10 degrees;
8. Passive Range of Motion at least 0 degrees ankle dorsiflexion in subtalar neutral or with FES

Exclusion Criteria:

1. A major, active, coexistent medical, neurological (apart from stroke) or psychiatric disease (apart from stroke), including alcoholism or dementia, orthopedic injuries, that substantially affects gait. **Because old orthopedic injuries may or may not affect gait, at the discretion of the site's study PI, exclusion criterion #2 related to orthopedic injuries can be waived if the injury was not on the stroke affected side and the joint/muscles are back to normal motor and range of motion function.
2. A major medical disorder that substantially reduces the likelihood that a subject will be able to comply with all study procedures or safely complete study procedures. This includes, but not limited to documented serious cardiac conditions, serious pulmonary conditions, legal blindness, end stage renal or liver disease, pulmonary embolism or deep venous thrombosis.
3. Resting systolic blood pressure above 170, diastolic blood pressure above 100 at screening and baseline evaluations
4. Implanted electronic device (e.g. pacemaker) or skull metallic implants (e.g. cranioplasty plate covering the leg motor area);
5. Deficits in communication that interfere with reasonable study participation: language or attention impairment (score>1 on NIH Stroke Scale items 9 and 11, respectively)
6. Significant cognitive impairment, defined as Montreal Cognitive Assessment score < 22 (For those with aphasia: **Because Montreal Cognitive Assessment scores may be difficult to interpret for patients with aphasia, at the discretion of the site's study PI, exclusion criterion #5 ("MoCA score cannot be <22") can be waived)
7. A new symptomatic stroke occurs apart from the index stroke during the screening process and prior to randomization
8. Life expectancy < 6 months
9. Skin breakdown over electrical stimulation sites;
10. Received chemical denervation (eg Botox) to legs in the preceding 6 months, or expectation that chemical denervation will be administered to the leg prior to expected completion of the study
11. Unable or unwilling to perform study procedures/therapy, or expectation of non-compliance with study procedures/therapy
12. Pregnancy;
13. Significant pain (visual analog scale >4), chest pain, or shortness of breath with walking.
14. Receiving any outside concurrent physical therapy involving the lower extremities after enrollment in the study up to 1 month post treatment
15. Any general medical condition and psychosocial situation that substantially interferes with reasonable participate in study appointments
16. Non-English speaking, such that subject does not speak sufficient English to comply with study procedures
17. Concurrent enrollment in another investigational interventional study
18. Severe depression, defined as Geriatric Depression Scale Score >11: **Because Geriatric Depression scale scores may be difficult to interpret for some patients, at the discretion of the site's study PI, exclusion criterion #17 ("Geriatric Depression score cannot be >11") can be waived)
19. Concurrent use of FES orthosis for gait.
20. A new symptomatic stroke occurs apart from the index stroke during the screening process and prior to randomization

    If TMS Eligible (note that potential subjects who do not qualify for TMS will not be excluded from the main study, they will only be excluded from undergoing TMS procedures):
21. TMS: Metallic hardware on the scalp (e.g. vascular clips or cranioplasty mesh)
22. TMS: Implanted medication pumps, intracardiac line, or central venous catheter
23. TMS: History of cortical stroke or other cortical lesion such as brain tumor
24. TMS: Prior diagnosis of seizure or epilepsy
25. TMS: Any electrical, mechanical, or magnetic implants
26. TMS: History of neurosurgery
27. TMS: uncontrolled Migraine headaches
28. TMS: Any current medications that affect seizure threshold such as tricyclic antidepressants and neuroleptics
29. TMS: Unstable medical conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine - Sue & Bill Gross Stem Cell Research Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biswas P, Dodakian L, Wang PT, Johnson CA, See J, Chan V, Chou C, Lazouras W, McKenzie AL, Reinkensmeyer DJ, Nguyen DV, Cramer SC, Do AH, Nenadic Z. A single-center, assessor-blinded, randomized controlled clinical trial to test the safety and efficacy of a novel brain-computer interface controlled functional electrical stimulation (BCI-FES) intervention for gait rehabilitation in the chronic stroke population. BMC Neurol. 2024 Jun 13;24(1):200. doi: 10.1186/s12883-024-03710-3. PMID 38872109

RESULTS

PARTICIPANT FLOW:
Groups:
- BCI-FES Dorsiflexion Therapy With Physiotherapy: Subjects will undergo placement of an EEG cap using standard technique connected to our custom BCI system. Subjects will provide 5 min of training EEG data as they engage in alternating epochs of idling and attempted foot dorsiflexion (of the paretic side). In the online phase, the subjects will perform ~10 BCI-FES runs (5 min/run). A total of 12 sessions will be performed at a rate of 3x/week (over 4 weeks). Each BCI-FES therapy session will be followed by 1 hour of conventional physiotherapy.
  Conventional Physical Therapy: This will consist of a standardized regimen of activities typical of conventional post-stroke gait therapy, including passive/active range of motion exercises (to reduce/prevent excessive plantarflexor contractures), lower-extremity muscle strengthening, and a progression from treadmill to overground walking exercises.
Period: Overall Study
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Started | 32 | 30
Completed | 29 | 26
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.03 (10.54) | 58.30 (12.85) | 59.19 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 24 | 13 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 18 | 17 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 26 | 22 | 48
  Unknown or Not Reported | 0 | 0 | 0
Gait Velocity [Mean (Standard Deviation); unit: m/s] | 0.38 (0.21) | 0.38 (0.26) | 0.38 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity
Description: Gait velocity will be assessed by measuring the time to traverse the middle 6 m of a 10-m walkway (5 repetitions/assessment). Scores are reported in meters/second with higher scores indicating better function.
Time Frame: Baseline to End of Therapy (4 weeks after initiation of therapy)
Population: Difference due to dropouts.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Number analyzed (Participants) | 32 | 30
m/s
  Baseline | 0.38 (0.21) | 0.38 (0.26)
  End of Therapy: number analyzed (Participants) | 29 | 26
  End of Therapy | 0.46 (0.23) | 0.45 (0.34)

2. Secondary Outcome: Dorsiflexion Range of Motion
Description: The paretic foot will be placed in a dangling, subtalar neutral position idling, while the tibia is perpendicular to the ground and the femur horizontal to the ground. A goniometer will be used to measure the maximum dorsiflexion angle, in degrees. 0 degrees indicates a neutral ankle position (foot horizontal to the ground, while tibia is perpendicular to the ground). Positive degrees indicate a maximum dorsiflexion angle above the neutral position, while negative degrees indicates a maximum angle below the neutral position (a larger, more positive measure indicates higher function).
Time Frame: Baseline and end of therapy (4 weeks after initiation of therapy)
Population: Difference due to dropouts
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Number analyzed (Participants) | 32 | 30
degrees
  Baseline | -12.54 (13.78) | -16.67 (15.78)
  End of Therapy: number analyzed (Participants) | 29 | 26
  End of Therapy | -10.05 (13.07) | -13.94 (15.74)

3. Secondary Outcome: Gait Endurance (Six Minute Walk Test: 6MWT)
Description: The distance walked over 6 minutes. Score is reported in meters and higher score indicates better function.
Time Frame: Baseline to End of Therapy (4 weeks after initiation of therapy)
Population: Difference due to drop outs.
Measure: Mean (Standard Deviation); unit: m
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Number analyzed (Participants) | 32 | 30
m
  Baseline | 101.08 (57.16) | 105.74 (75.60)
  End of Therapy: number analyzed (Participants) | 29 | 26
  End of Therapy | 118.19 (60.91) | 118.83 (85.38)

4. Secondary Outcome: Fall Frequency
Description: Rate of falls experienced by subjects
Time Frame: Baseline to End of Therapy (4 weeks after initiation of therapy)
Population: Difference due to drop outs.
Measure: Mean (Standard Deviation); unit: falls/week
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Number analyzed (Participants) | 32 | 30
falls/week
  Baseline | 0.11 (0.32) | 0.08 (0.27)
  End of Therapy: number analyzed (Participants) | 29 | 26
  End of Therapy | 0 (0) | 0 (0)

5. Secondary Outcome: EEG Map (Electroencephalogram)
Description: Subjects will undergo 64-channel EEG recording as they engage in 100 alternating 10-s long epochs of idling and attempted dorsiflexion. The EEG modulation, defined as the change in alpha (8-12 Hz) and beta (13-30 Hz) band power during attempted dorsiflexion (compared to idling) will be calculated and averaged over all epochs and across all channels. Change in EEG alpha and beta band power will be express as percentage with respect to the idle state. Specifically, the change in the Channel Cz will be reported given its primary salience to attempted dorsiflexion.
Time Frame: Baseline to End of Therapy (4 weeks after initiation of therapy)
Population: Difference in subjects due to dropouts.
Measure: Mean (Standard Deviation); unit: % of EEG alpha/beta power change
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
Number analyzed (Participants) | 32 | 30
% of EEG alpha/beta power change
  Baseline | -31.73 (18.55) | -39.48 (18.84)
  End of Therapy: number analyzed (Participants) | 29 | 26
  End of Therapy | -38.74 (25.10) | -36.33 (22.10)

ADVERSE EVENTS:
Time Frame: Baseline to End of 3-month post intervention follow up
Arm/Group | BCI-FES Dorsiflexion Therapy With Physiotherapy | Dose-and Intensity-matched Physiotherapy
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 7/32 | 3/30
Other Adverse Events (participants affected / at risk) | 3/32 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCI-FES Dorsiflexion Therapy With Physiotherapy (N=32) | Dose-and Intensity-matched Physiotherapy (N=30)
Severe adverse events (unrelated to study procedures) (Nervous system disorders) | 1 | 2
Falls with injury (unrelated to study procedures) (General disorders) | 2 | 0
Cardiac events (Cardiac disorders) | 3 | 1 — Deemed unrelated to study procedures
Orthopedic Injuries (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCI-FES Dorsiflexion Therapy With Physiotherapy (N=32) | Dose-and Intensity-matched Physiotherapy (N=30)
Pain (General disorders) | 2 | 0
Orthopedic Injury (Musculoskeletal and connective tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT04279067/Prot_SAP_000.pdf